CLINICAL TRIAL: NCT07196033
Title: Asian Gynecological Brachytherapy Registry in Cervical Cancer
Acronym: AGBR-FERN-Gyn
Status: Recruiting | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Chiang Mai University, Thailand (Unknown); Mahidol University (Other); Gunma University (Other); Juntendo University (Other)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Dr. Supriya Chopra, Tata Memorial Hospital
Other Study IDs: 901113
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Stage IIIA Cervical Cancer FIGO 2018; Stage IIIB Cervical Cancer FIGO 2018; Stage IVA Cervical Cancer FIGO 2018; Stage IB Cervical Cancer FIGO 2018; Stage IIA Cervical Cancer FIGO 2018; Stage IIB Cervical Cancer FIGO 2018
Keywords: Definitive chemo-radiation; Brachytherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gynecological cancer poses as significant public health issue, especially in Asian countries, where it is a leading cause of cancer-related deaths among women. Cervical cancer accounts for around 311,000 deaths annually, with over 85% occurring in low- and middle-income nations, primarily in Asia. Factors contributing to this burden include limited access to preventive care, inadequate screening, high rates of human papillomavirus infection, and cultural barriers that delay medical attention.

For patients with advanced cervical cancer, the standard treatment involves external beam radiation therapy along with chemotherapy followed by internal radiation, known as Brachytherapy. This technique uses unique set of devices placed internally at the tumor sitegiving localized radiation to the residual tumor tissue. While advanced brachytherapy techniques have been developed and practiced in Europe and American countries yielding excellent clinical outcomes, there is insufficient data on the use and results of such advanced brachytherapy techniques in Asian populations, leading to a lack of standardized practices.

To address these issues, the Asian Gynecological Brachytherapy Registry (ABGR) has been established as a collaborative platform for data collection and analysis on the use of Brachytherapy techniques. This registry aims to consolidate information from various healthcare settings across Asia, enhancing understanding of cervical cancer's epidemiology, evaluating treatment effectiveness, and identifying areas for improvement in patient care.

DETAILED DESCRIPTION:
The registry will follow a retrospective cohort study design by including consecutive patients treated in participating institutions over a 12-month period. It encompasses patients receiving various levels of brachytherapy, including 2D to 3D modalities, and considers different imaging techniques for treatment planning. Contouring variability and patient demographics are also accounted to ensure a comprehensive understanding of real-world application. With a target enrolment of 1,000 patients across multiple centres in FARO member countries, the AGBR aims to capture diverse patient environments and institutional practices. Through this collaborative effort, it seeks to report on different brachytherapy utilization patterns, clinical outcomes, and factors influencing treatment decisions and disparities. Additionally, information related to external radiation, administration of concurrent chemotherapy and overall treatment time will also be captured. Taken together these 3 components and timely administration of treatment constitute pillars of successful and effective treatment for cervix cancer. Administratively, data handling and storage protocols built in protocol will safeguard patient privacy and data integrity. Monitoring and quality assurance processes ensure data completeness and accuracy, while a publication policy promotes transparent dissemination of research findings, prioritizing multi-institutional collaborations and publishing in this domain from Asia.In conclusion, the AGBR once completed will represent a collaborative effort to address the variations in cervical cancer treatment in Asia and provide baseline data for future prospective work.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with FIGO 2018 stage IB-IVA cervical cancer with squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma histological subtype.
* Planned for treatment with definitive chemo-radiation and brachytherapy. (X- ray,CT, CT-Ultrasound or MRI based).

Exclusion Criteria:

* Neuroendocrine cancer of the cervix or other rare histology subtypes.
* Patients with metastatic cervix cancer and not planned for radical doses of pelvic RT/brachytherapy may be excluded.
* Patients undergoing postoperative RT or RT for recurrent disease should be excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is diagnosed with FIGO 2018 stage IB-IVA cervical cancer with squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma histological subtype and have undergone treatment with definitive chemo-radiation and brachytherapy (X-ray, CT, CT-Ultrasound or MRI based) for cervical cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-05-20 (Estimated)

PRIMARY OUTCOMES:
Recording and reporting the prevalent practices of cervical cancer brachytherapy in the management of cervical cancer in FARO member countries and report outcomes in reference to techniques utilised. | 3 years

SECONDARY OUTCOMES:
To record and report techniques utilised for external radiation and report outcomes in reference to EBRT techniques and prescription. | 3 years
To report utilisation rates of concurrent chemotherapy and report outcomes in reference to cumulative cisplatin dose delivered. | 3 years
. To record and report on prevalent brachytherapy fractionation regimes across participating sites. | 3 years
To record and report on overall treatment times for the management of cervical cancer. | 3 years
To report 2-yearlocal control, regional control and disease-free survival in reference to primary and nodal dose and chemotherapy dose in different subcohorts of cervical cancer. | 3 years
To report 2-year gastrointestinal, genitourinary, hematological and vaginal adverse events with use of radiation and brachytherapy using CTCAE version 5.0 | 3 years

CONTACTS AND LOCATIONS:
Locations (5):
- Tata Memorial Center, Mumbai, Maharashtra, India
- Japan (2):
  - Gunma University, Maebashi, Japan
  - Juntendo University, Tokyo, Japan
- Thailand (2):
  - Mahidol University, Bangkok, Thailand
  - Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hande V, Chopra S, Polo A, Mittal P, Kohle S, Ghadi Y, Mulani J, Gupta A, Kinhikar R, Agarwal JP. Transitioning India to advanced image based adaptive brachytherapy: a national impact analysis of upgrading National Cancer Grid cervix cancer guidelines. Lancet Reg Health Southeast Asia. 2023 Jun 6;16:100218. doi: 10.1016/j.lansea.2023.100218. eCollection 2023 Sep. PMID 37694176
- [Background] Tharavichitkul E, Mayurasakorn S, Lorvidhaya V, Sukthomya V, Wanwilairat S, Lookaew S, Pukanhaphan N, Chitapanarux I, Galalae R. Preliminary results of conformal computed tomography (CT)-based intracavitary brachytherapy (ICBT) for locally advanced cervical cancer: a single institution's experience. J Radiat Res. 2011;52(5):634-40. doi: 10.1269/jrr.10154. PMID 21952319
- [Background] Mittal P, Chopra S, Pant S, Mahantshetty U, Engineer R, Ghosh J, Gupta S, Ghadi Y, Menachery S, Swamidas J, Gurram L, Shrivastava SK. Standard Chemoradiation and Conventional Brachytherapy for Locally Advanced Cervical Cancer: Is It Still Applicable in the Era of Magnetic Resonance-Based Brachytherapy? J Glob Oncol. 2018 Jul;4:1-9. doi: 10.1200/JGO.18.00028. PMID 30085892
- [Background] Mahantshetty U, Krishnatry R, Hande V, Jamema S, Ghadi Y, Engineer R, Chopra S, Gurram L, Deshpande D, Shrviastava S. Magnetic Resonance Image Guided Adaptive Brachytherapy in Locally Advanced Cervical Cancer: An Experience From a Tertiary Cancer Center in a Low and Middle Income Countries Setting. Int J Radiat Oncol Biol Phys. 2017 Nov 1;99(3):608-617. doi: 10.1016/j.ijrobp.2017.06.010. Epub 2017 Jun 20. PMID 29280456
- [Background] Murakami N, Ando K, Murata M, Murata K, Ohno T, Aoshika T, Kato S, Okonogi N, Saito AI, Kim JY, Yoshioka Y, Sekii S, Tsujino K, Lowanichkiattikul C, Pattaranutaporn P, Kaneyasu Y, Nakagawa T, Watanabe M, Uno T, Umezawa R, Jingu K, Kanemoto A, Wakatsuki M, Shirai K, Igaki H, Itami J. An Asian multi-national multi-institutional retrospective study comparing intracavitary versus the hybrid of intracavitary and interstitial brachytherapy for locally advanced uterine cervical carcinoma. J Radiat Res. 2022 May 18;63(3):412-427. doi: 10.1093/jrr/rrac014. PMID 35446962
- [Background] Potter R, Tanderup K, Schmid MP, Jurgenliemk-Schulz I, Haie-Meder C, Fokdal LU, Sturdza AE, Hoskin P, Mahantshetty U, Segedin B, Bruheim K, Huang F, Rai B, Cooper R, van der Steen-Banasik E, Van Limbergen E, Pieters BR, Tan LT, Nout RA, De Leeuw AAC, Ristl R, Petric P, Nesvacil N, Kirchheiner K, Kirisits C, Lindegaard JC; EMBRACE Collaborative Group. MRI-guided adaptive brachytherapy in locally advanced cervical cancer (EMBRACE-I): a multicentre prospective cohort study. Lancet Oncol. 2021 Apr;22(4):538-547. doi: 10.1016/S1470-2045(20)30753-1. PMID 33794207
- [Background] Tharavichitkul E, Sivasomboon C, Wanwilairat S, Lorvidhaya V, Sukthomya V, Chakrabhandu S, Lookkaew S, Chitapanarux I, Galalae R. Preliminary results of MRI-guided brachytherapy in cervical carcinoma: the Chiangmai University experience. J Radiat Res. 2012;53(2):313-8. doi: 10.1269/jrr.11107. Epub 2012 Jan 21. PMID 22277978
- [Background] Tharavichitkul E, Jia-Mahasap B, Muangwong P, Chakrabandhu S, Klunklin P, Onchan W, Tippanya D, Nobnop W, Watcharawipha A, Kittidachanan K, Galalae RM, Chitapanarux I. Survival outcome of cervical cancer patients treated by image-guided brachytherapy: a 'real world' single center experience in Thailand from 2008 to 2018. J Radiat Res. 2022 Jul 19;63(4):657-665. doi: 10.1093/jrr/rrac025. PMID 35719089
- [Background] Singh D, Vignat J, Lorenzoni V, Eslahi M, Ginsburg O, Lauby-Secretan B, Arbyn M, Basu P, Bray F, Vaccarella S. Global estimates of incidence and mortality of cervical cancer in 2020: a baseline analysis of the WHO Global Cervical Cancer Elimination Initiative. Lancet Glob Health. 2023 Feb;11(2):e197-e206. doi: 10.1016/S2214-109X(22)00501-0. Epub 2022 Dec 14. PMID 36528031
- [Background] Schmid MP, Lindegaard JC, Mahantshetty U, Tanderup K, Jurgenliemk-Schulz I, Haie-Meder C, Fokdal LU, Sturdza A, Hoskin P, Segedin B, Bruheim K, Huang F, Rai B, Cooper R, van der Steen-Banasik E, Van Limbergen E, Pieters BR, Petric P, Ramazanova D, Ristl R, Kannan S, Hawaldar R, Ecker S, Kirchheiner K, Tan LT, Nout R, Nesvacil N, de Leeuw A, Potter R, Kirisits C; EMBRACE Collaborative Group. Risk Factors for Local Failure Following Chemoradiation and Magnetic Resonance Image-Guided Brachytherapy in Locally Advanced Cervical Cancer: Results From the EMBRACE-I Study. J Clin Oncol. 2023 Apr 1;41(10):1933-1942. doi: 10.1200/JCO.22.01096. Epub 2023 Jan 4. PMID 36599120